CLINICAL TRIAL: NCT07194460
Title: Effects of Combined Exercise and Peripheral Magnetic Stimulation on Biopsychosocial Functional Impairments in Older Adults With Schizophrenia
Brief Title: Combined Exercise and PMS: Impact on Biopsychosocial Function in Older Adults With Schizophrenia
Acronym: PMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuntong Zhang (Other)
Responsible Party: Sponsor-Investigator, Yuntong Zhang, Graduate Student, School of Rehabilitation, Shanghai University of Medicine & Health Sciences, Shanghai University of Medicine and Health Sciences
Organization: Shanghai University of Medicine and Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YJYZD202406; 202503650102197808083517 (Other: Clinical Research Ethics Committee, Shanghai University of Medicine & Health Sciences (SUMHS))
Record Dates: First submitted 2025-09-05; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia Patients
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study employs a triple-blind design. Patients, researchers, and data analysts are all blinded to the group assignments (treatment or control group) throughout the study. The randomization process is managed by an independent third party, and outcome data analysis is conducted by researchers who are unaware of group allocations. This ensures the minimization of bias during the trial and data interpretation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Peripheral Magnetic Stimulation (PMS) treatment group (Experimental): Treatment will be administered using a Peripheral Magnetic Stimulation (PMS) device. The intervention involves directing magnetic fields to stimulate specific peripheral nerve regions to regulate neural activity and improve symptoms.
  Interventions: Device: Peripheral Magnetic Stimulation (PMS)
- Sham control group (Sham Comparator): The placebo group will undergo a treatment process similar to the PMS intervention group, but without actual peripheral magnetic stimulation. The intervention will simulate the PMS treatment process, using a sham device that resembles the PMS device in appearance, but without generating any magnetic or electric field stimulation.
  Interventions: Device: ham control group receiving PMS intervention
- Exercise (Experimental): This exercise prescription includes four phases. First, a 5-minute warm-up (no sandbags/resistance bands) with walking in place, ankle rotations, and shoulder movements to boost blood flow and prevent injuries. Next, 10-12 minutes of leg strength training: sandbags for half squats (strengthen thighs, hips, knees), calf raises (enhance calf strength and lower limb stability), and resistance bands for standing leg abductions (improve hip/outer thigh strength/coordination). Then, 8-10 minutes of neurocoordination training with sandbags/resistance bands: marching in place (better leg coordination/endurance), gait training (improve balance/neural coordination), and step turns (increase gait flexibility/body control). Finally, a 5-minute relaxation with leg/ankle stretches to reduce post-exercise soreness.
  Interventions: Other: Exercise
- PMS＋Exercise (Experimental): Following the completion of PMS, exercise training is randomly conducted.
  Interventions: Other: PMS＋Exercise
- PMS (Experimental): This PMS refers to the peripheral magnetic stimulation administered in Experiment 2, serving to distinguish it from that in Experiment 1.
  Interventions: Device: Peripheral Magnetic Stimulation (PMS)

INTERVENTIONS:
Device: Peripheral Magnetic Stimulation (PMS) — Treatment will be administered using a Peripheral Magnetic Stimulation (PMS) device. The intervention involves directing magnetic fields to stimulate specific peripheral nerve regions to regulate neural activity and improve symptoms.
  Arms: PMS; Peripheral Magnetic Stimulation (PMS) treatment group
Device: ham control group receiving PMS intervention — Identical to the experimental group in all procedures, except that no electrical stimulation is delivered.
  Arms: Sham control group
Other: Exercise — See previous sections
  Arms: Exercise
Other: PMS＋Exercise — See previous sections
  Arms: PMS＋Exercise

SUMMARY:
This project consists of two randomized parallel - group experiments targeting older adults with schizophrenia, aiming to evaluate the therapeutic effect of Peripheral Magnetic Stimulation (PMS).

Experiment 1 (Efficacy of PMS): During a 4 - week intervention period, participants are randomly assigned to receive active PMS or sham PMS. The primary objective is to determine whether PMS can reduce the clinical symptom burden and improve biopsychosocial functioning compared with sham stimulation through electroencephalogram (EEG) signal acquisition and evaluation. Secondary objectives include the effects on cognition, mood, sleep, and health - related quality of life, as well as safety and tolerability (adverse events monitoring).

Experiment 2 (Comparison of Intervention Effects): The subjects are randomly divided into three groups: exercise combined with PMS group, PMS alone group, and exercise alone group. Each group is arranged by relevant professionals to carry out the corresponding intervention for 4 weeks. The main purpose is to examine the differences in the effects of the three intervention methods (exercise combined with PMS, PMS alone, and exercise alone) in improving patients' conditions, including the impact on exercise - related physical performance, functional mobility, etc. Secondary objectives include the impact on overall function and quality of life, along with safety monitoring.

In both experiments, outcome indicators are measured from baseline to post - intervention (and, where feasible, short - term follow - up) by assessors who are blinded to group allocation using appropriate tools. It is hypothesized that in Experiment 1, PMS will be superior to sham stimulation; in Experiment 2, the effect of exercise combined with PMS in improving patients' motor and related functions will be better than that of PMS alone or exercise alone, which supports PMS as a scalable auxiliary means for the rehabilitation of this population.

DETAILED DESCRIPTION:
Project Experimental Protocol (Revised Version) This project consists of two randomized parallel-group experiments involving older adults with schizophrenia, aiming to evaluate the therapeutic effects of Peripheral Magnetic Stimulation (PMS) and its potential to enhance exercise-related benefits. The rationale for this project is based on evidence that peripheral neuromuscular stimulation can modulate sensorimotor integration and functional mobility, while being well-tolerated in older populations.

Experiment 1 (Efficacy of PMS) Participants are randomly assigned to either the active PMS group or the sham PMS group, with interventions administered over several weeks in addition to standard care. Both participants and outcome assessors are blinded, and device operators are kept separate from assessors. PMS parameters, treatment protocols, and device details are specified in the "Interventions" section.

Outcome measures are collected at baseline and post-intervention (with short-term follow-up when feasible) using validated clinical scales, functional assessment tools, and patient-reported instruments. Additionally, electroencephalographic (EEG) signals are recorded to generate spectrograms, brain topographic maps, and brain functional connectivity maps. Specific analyses include: ① Observing changes in EEG energy across different frequency bands (e.g., alpha, beta, theta waves) via spectrograms to determine PMS-induced regulatory effects on brain electrical activity rhythms; ② Identifying regions of abnormal EEG activity using brain topographic maps to pinpoint core brain functional areas (e.g., sensorimotor cortex, prefrontal lobe) potentially affected by PMS; ③ Analyzing alterations in connectivity strength between brain regions (e.g., frontal-parietal, intrahemispheric) through functional connectivity maps to explore PMS-mediated modulation of neural circuit connectivity, thereby providing neurophysiological evidence for the mechanisms underlying PMS efficacy. Safety is monitored during each session in accordance with predefined termination criteria.

Experiment 2 (Enhancement of Exercise Benefits) This independent randomized trial randomly assigns participants to three groups: exercise combined with PMS group, PMS alone group, and exercise alone group, with each group receiving interventions for several weeks. The exercise combined with PMS group and the exercise alone group follow the same standardized, dose-matched exercise protocol, while the exercise combined with PMS group and the PMS alone group use consistent PMS intervention parameters. Outcome assessors are blinded, and therapists responsible for exercise instruction strictly adhere to uniform operational protocols across all three groups.

The core objective is to compare the efficacy differences among the three interventions, with key assessment indicators including: ① **Palm-held ultrasound measurement: Targeting key lower limb muscles (e.g., quadriceps femoris, gastrocnemius muscle), palm-held ultrasound is used to detect muscle thickness and echo intensity to evaluate intervention-induced improvements in muscle structure and quality; ② 6-minute walk test: Measuring the maximum distance walked by participants in 6 minutes to assess aerobic endurance and exercise endurance; ③ Sit-to-stand test: Recording the time/number of repetitions for participants to stand up from a seated position and sit back down to evaluate lower limb muscle strength, balance ability, and functional mobility; ④ Positive and Negative Syndrome Scale (PANSS) scores: Quantifying improvements in participants' psychiatric symptoms across three dimensions (positive symptoms, negative symptoms, general psychopathology). Other assessment domains (e.g., cognition, sleep, health-related quality of life) are consistent with those in Experiment 1. Participant adherence to interventions is enhanced through structured appointment reminders, intervention logs, and regular follow-ups.

Common Methods for Both Experiments

1. Randomization and Group Allocation**: Random sequences are computer-generated with concealed allocation. Stratification factors such as age, disease duration, and baseline motor ability may be incorporated as needed to reduce inter-group confounding.
2. Statistical Analysis： Analyses follow the intention-to-treat principle, using mixed-effects models to estimate group-by-time interaction effects and evaluate time-dependent impacts of interventions on outcomes. If model assumptions (e.g., normality, homoscedasticity) are violated, nonparametric tests (e.g., Wilcoxon rank-sum test) are used as alternatives. Multiple testing errors for confirmatory endpoints (e.g., PANSS scores, 6-minute walk distance, palm-held ultrasound-derived muscle thickness indicators) are controlled using the Holm-Bonferroni method, while the false discovery rate (FDR) method is applied to exploratory endpoints (e.g., EEG-derived metrics).
3. Data Processing: Missing data are handled using multiple imputation (generating 5-10 complete datasets), with sensitivity analyses of per-protocol populations to verify result stability. Data quality is ensured through assessor training (including PANSS rater consistency testing, standardized training for EEG data processing, and training on consistent operation of palm-held ultrasound), development of standard operating procedures (SOPs), and implementation of data range audits (e.g., excluding outliers beyond reasonable physiological ranges).
4. Ethical and Safety Oversight: The Institutional Review Board (IRB) provides full supervision, and intervention protocols require ethical approval before implementation. Adverse events (e.g., local skin irritation, dizziness) are recorded during each visit, classified by severity, and regularly submitted to the IRB for review.

To avoid redundancy, specific timelines for outcome measurement (e.g., EEG recording schedules, PANSS assessment frequency, palm-held ultrasound testing times), inclusion/exclusion criteria, sample size calculations, detailed study procedures, and PMS device parameters are described in their dedicated Patient-Reported Outcomes (PRO) fields/documents.

ELIGIBILITY:
# Eligibility Criteria

* Inclusion Criteria:

  * Participants must be aged ≥60 years.
  * Diagnosis of schizophrenia based on the International Classification of Diseases - 10th Edition (ICD-10) or Diagnostic and Statistical Manual of Mental Disorders - 5th Edition (DSM-5).
  * Diagnosis must be made for ≥6 months, with clinical manifestations of schizophrenia (e.g., hallucinations, delusions, thought disorder, etc.).
  * No history of severe acute psychiatric episodes or hospitalizations within the last 3 months prior to enrollment.
  * Symptoms must be controllable, with no reliance on acute psychiatric intervention.
  * Participants must be able to understand the study's purpose and procedures and provide written informed consent. If the participant is unable to provide full informed consent (e.g., due to severe cognitive impairment), informed consent must be obtained from a legal guardian.
* Exclusion Criteria:

  * Schizoaffective disorder or bipolar disorder with psychosis.
  * Elderly individuals with multiple chronic diseases but who still maintain good functional status and quality of life.
  * Presence of severe cardiovascular diseases, liver or kidney dysfunction, cerebrovascular diseases, or other physical conditions that may affect treatment.
  * Patients with contraindications to peripheral magnetic stimulation (PMS) treatment or EEG.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-28 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) score | After baseline assessment, participants will undergo either Peripheral Magnetic Stimulation (PMS) or exercise intervention, followed by follow-up assessments at Week 4 and Week 8.
  Positive and Negative Syndrome Scale (PANSS) Score
  Description: A 30-item scale assessing positive symptoms, negative symptoms, and general symptoms.
  Unit of Measure: Score (range 30-210)
resting-state electroencephalography (resting-state EEG) | Assessed at baseline (pre-intervention) and immediately post-intervention (within 30 minutes of the final session).
  Resting-State Electroencephalography (EEG)
  Description: EEG data collection and analysis, including 5-band power (δ, θ, α, β, γ) and brain connectivity.
  Unit of Measure: Microvolts squared per Hertz (μV²/Hz) for power bands, correlation coefficient for brain connectivity.
6-minute walk test | After baseline assessment, participants will undergo either Peripheral Magnetic Stimulation (PMS) or exercise intervention, followed by follow-up assessments at Week 4 and Week8 .
  6-Minute Walk Test (6MWT)
  Description: A standardized test measuring the distance walked in 6 minutes.
  Unit of Measure: Distance (meters)

SECONDARY OUTCOMES:
muscle mass index | Assessed at baseline (pre-intervention), at Week 4 follow-up, and at Week 8 follow-up
  Muscle Mass Index (using Palm-Held Ultrasound)
  Description: Measurement of muscle thickness and echo intensity at specific muscle sites.
  Unit of Measure:
  Muscle Thickness (millimeters, mm)
  Echo Intensity (decibels, dB)
Sit-to-Stand Test | Assessed at baseline (pre-intervention), at Week 4 follow-up, and at Week 8 follow-up
  Sit-to-Stand Test
  Description: Time to complete 5 sit-to-stand repetitions and the number of repetitions in 1 minute.
  Unit of Measure:
  Time (seconds) for 5 repetitions
  Repetitions per minute

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared, including baseline demographic characteristics (e.g., age, sex), primary and secondary outcome measures (e.g., Positive and Negative Syndrome Scale [PANSS] scores, muscle mass parameters from palm-sized ultrasound, resting-state EEG indices), intervention adherence, and adverse event data. Data will be provided in a format that does not contain any information that could directly identify participants.
Supporting Information: Study Protocol, ICF
Time Frame: after the article is published

DOCUMENTS (5):
  • Study Protocol: unchanged document (2024-05-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT07194460/Prot_000.pdf
  • Study Protocol and Statistical Analysis Plan: Align the update date with the ethics review date. (2025-05-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT07194460/Prot_SAP_001.pdf
  • Informed Consent Form: unchanged document (2025-05-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT07194460/ICF_002.pdf
  • Informed Consent Form: Align the update date with the ethics review date. (2025-05-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT07194460/ICF_003.pdf
  • Informed Consent Form: Align the update date with the ethics review date.（1） (2025-09-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT07194460/ICF_004.pdf